CLINICAL TRIAL: NCT06123910
Title: Effect of Bovine Colostrum Supplementation on Neutrophil Function in Recreational Athletes
Brief Title: Bovine Colostrum Supplementation in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigación en Alimentación y Desarrollo A.C. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: JHDEZ/CE/010-1/2018
Record Dates: First submitted 2023-10-16; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Innate Immunity
MeSH Terms: interventions — Refit milk powder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Colostrum bovine (Experimental): Subjets taking a colostrum supplement
  Interventions: Dietary Supplement: Colostrum bovine
- Placebo (Placebo Comparator): Subjets taking a commercial dairy product
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Colostrum bovine — Colostrum bovine supplements, 25 kcal per portion, containing 0.25 g fats, 2.0 g CHO and 3 g protein. Lactose reduced.
  Other Names: sovereign laboratories colostrum ld powder
  Arms: Colostrum bovine
Other: Placebo — Dairy comercial product. 25 kcal per portion, 1.3 g fats, 1.95 CHO and 1.3 protein. Lactose based.
  Other Names: Milk powder
  Arms: Placebo

SUMMARY:
32 recreational athletes who will attend to the Grand Marathon in the nort west of Mexico, event that will be held on December 2, 2018 or 21k Trail to be held in April 2019 will be invited to the study. Participants will be informed about the study procedures through a consent informed. Participants will be randomly divided into two groups, 16 in the intervention group and 16 in the comparison group. The participants will be recreational athletes between 18 and 60 years old. They must have athletic experience of at least 3 years. The participants considered will be those who perform vigorous physical activity per week according to the criteria of the short version IPAQ instrument. Smoking subjects with food intolerances and allergies, cardiovascular history will be excluded. Patients who have had a respiratory infection symptom in the last two weeks will not be able to participate in the study. Participants who are consuming some type of food supplement will be excluded.

Two 18 ml of blood samples will be taken from the vein of the forearm by venipuncture of each participant, using K2EDTA tubes after and before supplementation period. Blood samples were taken before a corporal, aerobic and nutritional evaluations.

CB supplementation will begin 4 weeks prior to competition events. One group will consume 20 g of bovine colostrum daily in solution with water. The second group will consume a placebo product with a nutritional composition similar to the group with the treatment of bovine colostrum. Both groups should take the supplement before breakfast with empty stomach.

DETAILED DESCRIPTION:
It is widely accepted that exercise provide important health benefits. However, vigorous or extenuate exercise can affect the correct function of the immune system. Athletes who perform extreme physical routines to improve their athletic performance can develop opportunistic infections. After 3 to 72 h of physical activity there is a phase called "open window for infection", which predispose to upper track respiratory infection (UTRI). URTI is the main cause of medical consultation in athletes with vigorous exercise practices.

Neutrophils are one of the most abundant leucocytes in blood; their phagocytic activity is essential to control bacterial infections. Recently, the interest in knowing the participation of these cells in the sport field is growing. Neutrophilia refers to a high concentration of neutrophils in blood, and this is a common condition after exercise. The controversial part is that vigorous exercise could limit some important functions, such as oxidative burst, degranulation and phagocytosis until 6 h after exercise. However, there are contradictory results in this topic.

To alleviate those immunological alterations in athletes, a nutritional intervention should be included. Bovine colostrum has been evaluated as a supplement due to its potential immunomodulatory properties. It improves immunological parameters in individuals who achieve prolonged exercise sessions, allowing URTI reduction. Bovine colostrum is a yellow aqueous compound secreted by cow mammary glands the first 72 h after partum. Bovine colostrum contains anti-microbial peptides, enzymes, immunoglobulins, cytokines, microRNA and growth factors, which are able to modulate the immune system, at local (intestinal) and systemic level. Due to these characteristics, bovine colostrum has been used to improve the immune response under different physiological conditions.

A study showed that bovine colostrum supplementation induces a CD89 expression pre-exercise, after 5 weeks supplementation with 10 g of bovine colostrum. This result is important, since CD89 is a membrane receptor in neutrophils that recognize antibody/antigen complexes to prime phagocytosis and degranulation. In other study, 3 weeks of bovine colostrum supplementation improved neutrophil degranulation 1 h post-exercise in athletes, after 2 h of physical exercise. Authors evaluated neutrophil oxidative burst post-exercise after bovine colostrum supplementation, but no effects were observed. However, these authors found better oxidative burst after 4 weeks bovine colostrum supplementation. At this time, the effect of bovine colostrum in phagocytosis activity is unknown.

Concerning the effects of bovine colostrum supplementation in the URTI incidence, the results are contradictory. Although, others found no benefit in the incidence of URTI after a bovine colostrum supplementation, other studies showed promising results. A retrospective analysis conducted in 2003 showed a reduction of athletes with URTI in the bovine colostrum supplementation group. Likewise, another study reported less episodes and duration of infections in physically active subjects. Other studies described a tendency to decrease the incidence of URTI in swimmers and cyclists.

Study Design

A total of 28 athletes attending the "Hermosillo Grand Marathon" (December 2, 2018) and/or the "Hermosillo Half Marathon" (March 2019) will be part of this study. In this randomized clinical trial, study subjects will be randomly divided in two groups, 14 in the intervention group (bovine colostrum supplementation) and 14 in the comparison group (placebo supplementation). The participants will be recreational athletes between 18 and 60 years old. They must have athletic experience of at least 3 years and have to perform a vigorous physical activity per week according to the criteria of the short version IPAQ instrument. Smoking subjects, with food intolerances, allergies or cardiovascular history will not be included. Athletes with respiratory infection symptoms two weeks before beginning the supplementation won't be part of this protocol. Participants who are consuming some other type of food supplement will not be included. This protocol is currently under evaluation of the Ethics Committee of our institution. Participants will be informed about the study procedures and will sign an informed consent.

Bovine colostrum supplementation will begin 4 weeks prior to the competition event. The intervention group will consume 20 g of bovine colostrum, divided into two doses of 10 g/day. The first dose will be before breakfast and the second before lunch. The comparison group will consume a placebo product.

Two blood samples (24 ml of each one) will be taken from the vein of the forearm of each participant, using tubes with EDTA. The first sample will be taken before the competitive event after 10 min of a sitting rest. The second sample will be obtained immediately at the end of the test with 3 minutes of sitting rest.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 years of training experience
* training for a half marathon competition
* No smokers
* Taking any kind of food supplements
* No alimentary allergies

Exclusion Criteria:

* Injuries
* not follow experimental indications
* cardiovascular disease
* treatment intolerances

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Neutrophil phagocytic capacity | Before and after 4 weeks of supplementation
  Percentage of phagocytic neutrophils
Monocytes phagocytic capacity | Before and after 4 weeks of supplementation
  Percentage of phagocytic monocytes
neutrophils producing reactive oxygen species | before and after 4 weeks of supplementation
  percentage of positive cells to fluorescence intensity by flow cytometry
neutrophils reactive oxygen species production intensity | Before and after 4 weeks of supplementation
  Mean intensity fluorescent by cells measured by flow cytometry
Monocytes producing reactive oxygen species | before and after 4 weeks of supplementation
  percentage of positive cells to fluorescence intensity by flow cytometry
Monocytes reactive oxygen species production intensity | Before and after 4 weeks of supplementation
  Mean intensity fluorescent by cells measured by flow cytometry
VO2Max | Before and after 4 weeks of supplementation
  Indicates participants aerobic condition (ml/kg/min)
Days presenting upper respiratory tract symptoms | During supplementation 4 weeks of supplementation
  Total of days that participants refers any kind of upper respiratory symptoms

SECONDARY OUTCOMES:
Weight | before and after 4 weeks of supplementation
  Weight in kilograms
Height | before and after 4 weeks of supplementation
  Height in meters
Body fat | before and after 4 weeks of supplementation
  Body fat percentage
Fat free mass | before and after 4 weeks of supplementation
  fat free mass percentage
Energy consumption | before, after 2 and 4 weeks of supplementation
  Measure of regular calories consumption in kcal by 24 h records method
Macronutrient consumption | before, after 2 weeks and 4 weeks of supplementation
  Measure of regular consumption of carbohydrates in grams, Protein in grams, fats in grams by 24 h records method

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Hernández, PhD, Principal Investigator — Centro de Investigación en Alimentación y Desarrollo A.C.
Locations (1):
- Centro de Investigación en Alimentación y Desarrollo, Hermosillo, Sonora, Mexico

REFERENCES:
- [Background] Hackney AC, Koltun KJ. The immune system and overtraining in athletes: clinical implications. Acta Clin Croat. 2012 Dec;51(4):633-41. PMID 23540172
- [Background] Li TL, Gleeson M. The effect of single and repeated bouts of prolonged cycling on leukocyte redistribution, neutrophil degranulation, IL-6, and plasma stress hormone responses. Int J Sport Nutr Exerc Metab. 2004 Oct;14(5):501-16. doi: 10.1123/ijsnem.14.5.501. PMID 15673097
- [Background] Peake J, Suzuki K. Neutrophil activation, antioxidant supplements and exercise-induced oxidative stress. Exerc Immunol Rev. 2004;10:129-41. PMID 15633591
- [Background] Tritto ACC, Amano MT, De Cillo ME, Oliveira VA, Mendes SH, Yoshioka C, Roschel H, Camara NOS, Gualano B, Artioli GG. Effect of rapid weight loss and glutamine supplementation on immunosuppression of combat athletes: a double-blind, placebo-controlled study. J Exerc Rehabil. 2018 Feb 26;14(1):83-92. doi: 10.12965/jer.1835154.577. eCollection 2018 Feb. PMID 29511657
- [Background] Bermon S, Castell LM, Calder PC, Bishop NC, Blomstrand E, Mooren FC, Kruger K, Kavazis AN, Quindry JC, Senchina DS, Nieman DC, Gleeson M, Pyne DB, Kitic CM, Close GL, Larson-Meyer DE, Marcos A, Meydani SN, Wu D, Walsh NP, Nagatomi R. Consensus Statement Immunonutrition and Exercise. Exerc Immunol Rev. 2017;23:8-50. PMID 28224969
- [Background] Jones AW, Thatcher R, March DS, Davison G. Influence of 4 weeks of bovine colostrum supplementation on neutrophil and mucosal immune responses to prolonged cycling. Scand J Med Sci Sports. 2015 Dec;25(6):788-96. doi: 10.1111/sms.12433. Epub 2015 Feb 28. PMID 25727914
- [Background] Shing CM, Peake J, Suzuki K, Okutsu M, Pereira R, Stevenson L, Jenkins DG, Coombes JS. Effects of bovine colostrum supplementation on immune variables in highly trained cyclists. J Appl Physiol (1985). 2007 Mar;102(3):1113-22. doi: 10.1152/japplphysiol.00553.2006. Epub 2006 Nov 9. PMID 17095643
- [Background] Rathe M, Muller K, Sangild PT, Husby S. Clinical applications of bovine colostrum therapy: a systematic review. Nutr Rev. 2014 Apr;72(4):237-54. doi: 10.1111/nure.12089. Epub 2014 Feb 26. PMID 24571383
- [Background] Crooks CV, Wall CR, Cross ML, Rutherfurd-Markwick KJ. The effect of bovine colostrum supplementation on salivary IgA in distance runners. Int J Sport Nutr Exerc Metab. 2006 Feb;16(1):47-64. doi: 10.1123/ijsnem.16.1.47. PMID 16676703
- [Result] Soligard T, Steffen K, Palmer D, Alonso JM, Bahr R, Lopes AD, Dvorak J, Grant ME, Meeuwisse W, Mountjoy M, Pena Costa LO, Salmina N, Budgett R, Engebretsen L. Sports injury and illness incidence in the Rio de Janeiro 2016 Olympic Summer Games: A prospective study of 11274 athletes from 207 countries. Br J Sports Med. 2017 Sep;51(17):1265-1271. doi: 10.1136/bjsports-2017-097956. Epub 2017 Jul 29. PMID 28756389
- [Result] Palmer-Green D, Elliott N. Sports injury and illness epidemiology: Great Britain Olympic Team (TeamGB) surveillance during the Sochi 2014 Winter Olympic Games. Br J Sports Med. 2015 Jan;49(1):25-9. doi: 10.1136/bjsports-2014-094206. Epub 2014 Nov 25. PMID 25425714
- [Result] McCarthy DA, Macdonald I, Grant M, Marbut M, Watling M, Nicholson S, Deeks JJ, Wade AJ, Perry JD. Studies on the immediate and delayed leucocytosis elicited by brief (30-min) strenuous exercise. Eur J Appl Physiol Occup Physiol. 1992;64(6):513-7. doi: 10.1007/BF00843760. PMID 1618188
- [Result] Davison G, Diment BC. Bovine colostrum supplementation attenuates the decrease of salivary lysozyme and enhances the recovery of neutrophil function after prolonged exercise. Br J Nutr. 2010 May;103(10):1425-32. doi: 10.1017/S0007114509993503. Epub 2009 Dec 24. PMID 20030905
- [Result] Pyne DB, Baker MS, Fricker PA, McDonald WA, Telford RD, Weidemann MJ. Effects of an intensive 12-wk training program by elite swimmers on neutrophil oxidative activity. Med Sci Sports Exerc. 1995 Apr;27(4):536-42. PMID 7791584
- [Result] Robson PJ, Blannin AK, Walsh NP, Castell LM, Gleeson M. Effects of exercise intensity, duration and recovery on in vitro neutrophil function in male athletes. Int J Sports Med. 1999 Feb;20(2):128-35. doi: 10.1055/s-2007-971106. PMID 10190775
- [Result] Santos VC, Levada-Pires AC, Alves SR, Pithon-Curi TC, Curi R, Cury-Boaventura MF. Changes in lymphocyte and neutrophil function induced by a marathon race. Cell Biochem Funct. 2013 Apr;31(3):237-43. doi: 10.1002/cbf.2877. Epub 2012 Sep 13. PMID 22972482
- [Result] Brinkworth GD, Buckley JD. Concentrated bovine colostrum protein supplementation reduces the incidence of self-reported symptoms of upper respiratory tract infection in adult males. Eur J Nutr. 2003 Aug;42(4):228-32. doi: 10.1007/s00394-003-0410-x. PMID 12923655
- [Result] Crooks C, Cross ML, Wall C, Ali A. Effect of bovine colostrum supplementation on respiratory tract mucosal defenses in swimmers. Int J Sport Nutr Exerc Metab. 2010 Jun;20(3):224-35. doi: 10.1123/ijsnem.20.3.224. PMID 20601740